CLINICAL TRIAL: NCT06461234
Title: Establishment of an Artificial Intelligence Multidimensional Early Warning Diagnostic and Prognostic Model of Pelvic Floor Rehabilitation Therapy in the Chinese Population: a Prospective Cohort Study.
Brief Title: Pelvic Floor Rehabilitation of Female Pelvic Floor Dysfunction
Status: Recruiting | Type: Observational
Sponsor: Mingfu Wu (Other)
Collaborators: Peking Union Medical College Hospital (Other); Peking University Third Hospital (Other); The Second Hospital of Shandong University (Other); Changsha Hospital for Maternal and Child Health Care (Other); Southwest Hospital, China (Other); Hangzhou Women's Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Mingfu Wu, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: 2024-S097
Record Dates: First submitted 2024-05-27; First posted 2024-06-14 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Pelvic Floor Disorders; Pelvic Organ Prolapse
Keywords: Pelvic Organ Prolapse; pelvic floor rehabilitation; pelvic floor muscle training; biofeedback electrical stimulation; magnetic stimulation
MeSH Terms: conditions — Pelvic Floor Disorders; Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- pelvic floor muscle training (PFMT): Control group
  Interventions: Behavioral: Pelvic floor muscle training
- pelvic floor biofeedback electrical stimulation: Observation Group 1
  Interventions: Other: Biofeedback electrical stimulation
- pelvic floor magnetic stimulation: Observation Group 2
  Interventions: Other: Magnetic Stimulation
- Magnetic stimulation combined with biofeedback electrical stimulation: Observation Group 3
  Interventions: Other: Magnetic stimulation combined with biofeedback electrical stimulation

INTERVENTIONS:
Behavioral: Pelvic floor muscle training — A therapist will instruct the patient to contract the anus, perineum as well as the urethra, until the patient masters the correct method.
  Groups: pelvic floor muscle training (PFMT)
Other: Biofeedback electrical stimulation — The therapist will place the electrodes of the instrument into the vagina, adjust the current value until the woman feels obvious contraction of the pelvic floor muscles but no pain, and instructs the patient to refer to the biofeedback mode for vaginal and anal contraction and relaxation.
  Groups: pelvic floor biofeedback electrical stimulation
Other: Magnetic Stimulation — The therapist will use the magnetic stimulator to intermittently stimulate the and adjust the stimulation intensity at any time according to the patient&#39;s condition, adjusting it until there is a clear sense of contraction and feel comfortable.
  Groups: pelvic floor magnetic stimulation
Other: Magnetic stimulation combined with biofeedback electrical stimulation — Pelvic floor magnetic stimulation for 30 minutes followed by biofeedback electrical stimulation.
  Groups: Magnetic stimulation combined with biofeedback electrical stimulation

SUMMARY:
The goal of this observational study is to learn about the therapeutic effects of different pelvic floor rehabilitation treatments, including pelvic floor muscle training , pelvic floor biofeedback electrical stimulation, and magnetic stimulation, in a population of Chinese patients with female pelvic floor dysfunction disorders. The study aims to find out the individualised pelvic floor rehabilitation treatment plan suitable for the Chinese population. The main question it aims to answer is:

1. Do patients with reduced pelvic floor muscle strength after childbirth, or patients with mild to moderate pelvic organ prolapse and symptomatic pelvic organ prolapse benefit from pelvic floor rehabilitation?
2. Is the combination of biofeedback electrical stimulation plus pelvic floor magnetic stimulation superior to single electrical stimulation, magnetic stimulation or pelvic floor muscle training?
3. Which pelvic floor rehabilitation therapy is most suitable for Chinese patients with female pelvic floor dysfunction?
4. What factors are early predictors of developing female pelvic floor dysfunction? And what factors can predict the prognostic status of patients treated with pelvic floor rehabilitation? Participants in the multicenter will be treated with different rehabilitation therapies, during which the researchers will collect clinical symptoms using the PFDI20 questionnaire, and POP-Q scores, pelvic floor muscle strength, and electromyography results from participants before, at the end of, and 3 months and 1 year after the end of treatment.

DETAILED DESCRIPTION:
This multicentre, prospective cohort study will be conducted at seven hospital-based pelvic floor health centres nationwide in China. Patients with pelvic floor dysfunctional disorders who are scheduled to undergo pelvic floor rehabilitation are included, including 1) postpartum pelvic floor muscle weakness, 2) mild-to-moderate pelvic organ prolapse (POP), and 3) POP in combination with dysfunction (bowel or bladder dysfunction) or POP in combination with lower urinary tract symptoms (overactive bladder syndrome, constipation, faecal incontinence).

Pelvic floor rehabilitation was performed in accordance with the clinical pathway based on patients' disease characteristics and individual conditions, during which baseline data were collected from patients who met the inclusion and exclusion criteria, as well as follow-up surveys at the end of the treatment, 3 months after the end of the treatment, and 12 months after the end of the treatment. The clinical data collected were used to determine the effectiveness of treatment and to summarise the effects of different rehabilitation programmes on the prognosis of postpartum and middle-aged and elderly PFD patients. The data were matched and compared with the patients' clinical symptoms, signs and auxiliary examinations, so as to optimise and determine the individualised and precise pelvic floor rehabilitation treatment plan.

ELIGIBILITY:
Inclusion Criteria:

1. knowledge of the study, voluntary enrolment in the study, and signing of informed consent;
2. postpartum pelvic floor weakness (pelvic floor muscle strength less than grade 3), or mild to moderate pelvic organ prolapse (POP-Q staging less than stage III), or pelvic organ prolapse combined with dysfunction (bowel or bladder dysfunction).

Exclusion Criteria:

1. history of comorbid serious medical or surgical illness;
2. comorbid psychiatric disorders;
3. contraindications to electrical and magnetic stimulation such as implanted pacemakers;
4. pelvic malignancy, acute genitourinary infection or vaginal bleeding, and genital tract malformation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is aimed at female patients with pelvic floor dysfunction. A large group of people are women who develop reduced pelvic floor muscle strength after childbirth; these women may not present with organic changes in the pelvic organs, but may present with symptoms such as unsatisfactory sexual behaviour and stress urinary incontinence as a result of weakened muscle strength. The other part of the population is patients with mild to moderate pelvic organ prolapse, where physical examination may reveal mild to moderate prolapse of the anterior vaginal wall, uterus, or posterior vaginal wall. If this group of patients had a combination of urinary and gastrointestinal symptoms, they could also be included in the study.
Sampling Method: Probability Sample
Enrollment: 1360 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
pelvic floor muscle strength | Baseline, 0 month and 3 months after pelvic floor rehabilitation treatment
  Pelvic floor muscle strength was assessed with reference to the Modified Oxford Muscle Strength Classification Method. Pelvic floor muscle strength was graded on a scale of 0-5: 0 for no contraction; 1 for tremor; 2 for slight contraction, with increased muscle strength but no lifting sensation; 3 for moderate contraction, with a sense of lifting of the posterior vaginal wall; 4 for good contraction, with a sense of lifting of the posterior vaginal wall against resistance; and 5 for strong contraction, with a sense of strong wrapping. The higher the grade, the better the pelvic floor strength.
pelvic floor electromyography | Baseline, 0 month and 3 months after pelvic floor rehabilitation.
  Pelvic floor electromyography is assessed by the pelvic floor surface electromyography analysis and biofeedback training system. EMG values and parameters regarding muscle contraction and relaxation will be recorded.

SECONDARY OUTCOMES:
POP-Q | Baseline, 0 month and 3 months after pelvic floor rehabilitation.
  The patient empties the bladder in a quiet state and is examined in the truncated position, the maximum degree of prolapse that can be achieved with a forceful downward breath-hold in the Valsalva manoeuvre.
PFDI-20 | Baseline, , 0 month, 3 months and 1 year after pelvic floor rehabilitation.
  Clinical symptoms are collected using the validated Chinese version of the international standardised questionnaire: PFDI-20, and patients are asked to select the answers that apply to their situation.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang AC, Wang YY, Chen MC. Single-blind, randomized trial of pelvic floor muscle training, biofeedback-assisted pelvic floor muscle training, and electrical stimulation in the management of overactive bladder. Urology. 2004 Jan;63(1):61-6. doi: 10.1016/j.urology.2003.08.047. PMID 14751349
- [Background] Terlikowski R, Dobrzycka B, Kinalski M, Kuryliszyn-Moskal A, Terlikowski SJ. Transvaginal electrical stimulation with surface-EMG biofeedback in managing stress urinary incontinence in women of premenopausal age: a double-blind, placebo-controlled, randomized clinical trial. Int Urogynecol J. 2013 Oct;24(10):1631-8. doi: 10.1007/s00192-013-2071-5. Epub 2013 Feb 27. PMID 23443345
- [Background] Feng F, Ashton-Miller JA, DeLancey JOL, Luo J. Feasibility of a deep learning-based method for automated localization of pelvic floor landmarks using stress MR images. Int Urogynecol J. 2021 Nov;32(11):3069-3075. doi: 10.1007/s00192-020-04626-5. Epub 2021 Jan 21. PMID 33475815
- [Background] Zhang L, Wang F. Evaluation of Nursing Effects of Pelvic Floor Muscle Rehabilitation Exercise on Gastrointestinal Tract Rectal Cancer Patients Receiving Anus-preserving Operation by Intelligent Algorithm-based Magnetic Resonance Imaging. Contrast Media Mol Imaging. 2022 May 19;2022:1613632. doi: 10.1155/2022/1613632. eCollection 2022. PMID 35655733
- [Background] Wang X, He D, Feng F, Ashton-Miller JA, DeLancey JOL, Luo J. Multi-label classification of pelvic organ prolapse using stress magnetic resonance imaging with deep learning. Int Urogynecol J. 2022 Oct;33(10):2869-2877. doi: 10.1007/s00192-021-05064-7. Epub 2022 Jan 27. PMID 35083500
- [Background] Nygaard I, Barber MD, Burgio KL, Kenton K, Meikle S, Schaffer J, Spino C, Whitehead WE, Wu J, Brody DJ; Pelvic Floor Disorders Network. Prevalence of symptomatic pelvic floor disorders in US women. JAMA. 2008 Sep 17;300(11):1311-6. doi: 10.1001/jama.300.11.1311. PMID 18799443
- [Background] Erekson EA, Fried TR, Martin DK, Rutherford TJ, Strohbehn K, Bynum JP. Frailty, cognitive impairment, and functional disability in older women with female pelvic floor dysfunction. Int Urogynecol J. 2015 Jun;26(6):823-30. doi: 10.1007/s00192-014-2596-2. Epub 2014 Dec 17. PMID 25516232
- [Background] Hong MK, Ding DC. Current Treatments for Female Pelvic Floor Dysfunctions. Gynecol Minim Invasive Ther. 2019 Oct 24;8(4):143-148. doi: 10.4103/GMIT.GMIT_7_19. eCollection 2019 Oct-Dec. PMID 31741838